CLINICAL TRIAL: NCT00820378
Title: Epidemiology of Aortic Dimensions in Patients With Clinically Evident Arterial Disease or Cardiovascular Risk Factors
Brief Title: The Epidemiology of Aortic Diameter in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Taizhou Hospital (Other)
Responsible Party: Jian-an Wang/Prof., Second Affiliated Hospital, College of Medicine, Zhejiang University
Other Study IDs: EPAD
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Vascular Disease; Diabetes; Hypertension; Hyperlipidemia
Keywords: Aortic dimension; Atherosclerosis; Vascular disease; Risk factors
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Hypertension; Hyperlipidemias; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- atherosclerosis: Patients With Clinically Evident Arterial Disease or Cardiovascular Risk Factors
  Interventions: Other: No special interventioin

INTERVENTIONS:
Other: No special interventioin — Comprehensive transthoracic M-mode, 2-dimensional, and Doppler echocardiographic studies will be performed using commercially available equipment. The aortic dimensions were assessed at end-diastole at the different levels:

SUMMARY:
Aortic aneurysms are the major disease processes affecting the aorta and becoming a relatively common cause of death because of rupture or dissection. The most common location for aneurysms is the infrarenal abdominal aorta, followed by the ascending thoracic aorta. Unlike coronary heart disease, the incidence of abdominal aortic aneurysm (AAA) in the United States and Europe has been increasing, and this increase may not be due to higher levels of screening for this condition alone. Aortic diameter is central to the diagnosis of aortic aneurysm. Furthermore, it was demonstrated that non-AAA patients with an enlarged diameter of the infrarenal aortic diameter are also at high risk for all-cause mortality. And aortic root dimension was associated with several coronary artery disease (CHD) risk factors and measures of subclinical disease and was predictive of incident congestive heart failure (CHF), stroke, cardiovascular disease (CVD) mortality, and all-cause mortality, but not of incident MI. Up to now, there are limited studies on the epidemiology of aortic diameter, especially in Chinese population.

DETAILED DESCRIPTION:
The purpose of this study was to analyze the size of the entire aorta at different anatomic levels in a large group of Chinese population with clinically evident arterial disease or cardiovascular risk factors to further explored the risk factors and potential alternative pathomechanisms for the development of aortic dilatation. Comprehensive transthoracic M-mode, 2-dimensional, and Doppler echocardiographic studies will be performed using commercially available equipment. The aortic dimensions were assessed at end-diastole at the different levels: (1) the annulus, (2) the mid-point of the sinuses of Valsalva, (3) the sinotubular junction, (4) the ascending aorta at the level of its largest diameter, (5) the transverse arch, (6) the descending aorta posterior to the left atrium, and (7) the abdominal aorta just distal to the origin of the renal arteries. The extension of dilation is defined as the number of dilated aortic segments. The relations among aortic dimensions and clinical characteristics will be assessed by multiple regression analysis. The current study was to determine the association of risk factors of CVD and atherosclerosis diseases with aortic dimension in Chinese patients with clinical event atherosclerotic disease or risk factors of atherosclerotic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 100 were referred to the hospital with a recent diagnosis of clinically evident arterial disease or a cardiovascular risk factor.

Exclusion Criteria:

* Those with connective tissue disease, congenital heart disease, cardiomyopathy, congestive heart failure,rheumatic arthritis, secondary causes of hypertension, or active cancer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population with clinically evident arterial disease or cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University; Li-jiang Tang, Principal Investigator — Taizhou Hospital, Wenzhou Medical College; Xiao-feng Chen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Zhao-xia Pu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xian-fang Lin, Principal Investigator — Taizhou Hospital, Wenzhou Medical College
Locations (2):
- China (2):
  - Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital, Wenzhou Medical College, Taizhou, Zhejiang